CLINICAL TRIAL: NCT01955096
Title: Fast Track Surgery With Laparoscopic-assisted Gastrectomy for Advanced Gastric
Brief Title: Fast Track Surgery With Laparoscopic-assisted Gastrectomy for Advanced Gastric Cancer: a Randomized Controlled Trial
Acronym: FTSlapAG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Quan Wang (Other)
Responsible Party: Sponsor-Investigator, Quan Wang, Deputy Director of General Surgery, The First Hospital of Jilin University
Organization: The First Hospital of Jilin University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2013-172; 2013-172 (Registry Identifier: Quan Wang)
Record Dates: First submitted 2013-09-25; First posted 2013-10-07 (Estimated); Last update posted 2013-10-09 (Estimated); Status verified 2013-10

CONDITIONS: Gastric Cancer
Keywords: fast-track surgery, laparoscopic gastrectomy
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- fast-track surgery (Experimental): The included patients will be randomly divided to two groups :30 that will undergo LAG with FTS rehabilitation programme and 31 that also will undergo LAG but receive conventional postoperative care.Laparoscopy-assisted gastrectomy will be carried out in this approach.There will be no difference in the surgical procedures of both groups.The criteria for discharge are: tolerance of solid diet, return of bowel habits and ability to walk on their own.
  Interventions: Procedure: fast-track surgery
- conventional postoperative care (Other): The included patients will be randomly divided to two groups :30 that will undergo LAG with FTS rehabilitation programme and 31 that also will undergo LAG but receive conventional postoperative care.Laparoscopy-assisted gastrectomy will be carried out in this approach.There will be no difference in the surgical procedures of both groups.The criteria for discharge are: tolerance of solid diet, return of bowel habits and ability to walk on their own.
  Interventions: Procedure: conventional postoperative care

INTERVENTIONS:
Procedure: fast-track surgery — The included patients will be randomly divided to two groups :30 that will undergo LAG with FTS rehabilitation programme and 31 that also will undergo LAG but receive conventional postoperative care.Laparoscopy-assisted gastrectomy will be carried out in this approach.There will be no difference in the surgical procedures of both groups.The criteria for discharge are: tolerance of solid diet, return of bowel habits and ability to walk on their own.
  Arms: fast-track surgery
Procedure: conventional postoperative care — The included patients will be randomly divided to two groups :30 that will undergo LAG with FTS rehabilitation programme and 31 that also will undergo LAG but receive conventional postoperative care.Laparoscopy-assisted gastrectomy will be carried out in this approach.There will be no difference in the surgical procedures of both groups.The criteria for discharge are: tolerance of solid diet, return of bowel habits and ability to walk on their own.
  Arms: conventional postoperative care

SUMMARY:
The purpose of this study is to to investigate the feasibility and safety of fast-track surgery when combined with laparoscopic-assisted gastrectomy for advanced gastric cancer patients.

DETAILED DESCRIPTION:
Methods: We designed a prospective randomized, controlled clinical trial then recruited 61 consecutive advanced gastric cancer patients. (Trial registration number: JLUFHC1722013) Further divide into a fast-track surgery group (n=30) and a conventional surgery group (n=31). Surgical technique in both groups is same laparoscopic-assisted gastrectomy with D2 lymphadenectomy. Compare outcomes includes length of hospital stay, return to normal diet and postoperative complications.Results: Recovery parameters such as the length of time to return to normal diet; to the first defection; start of ambulation time ;the mean hospital stay will be all less in patients assigned to the fast track surgery protocol compared with those in the conventional care programme. Conclusion: We will consider fast-track rehabilitation to be safe and feasible in advanced gastric cancer patients. Moreover, it will result in decreased hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of advanced gastric cancer, elective laparoscopic surgery and age under 75.

Exclusion Criteria:

* Patients with early gastric cancer, received neoadjuvant chemotherapy, had pyloric obstruction or with distant metastasis were excluded from the study.

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2010-09; Primary Completion 2012-09 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Ambulation time | within the first 30 days (plus or minus 3 days) after surgery
defection time | within the first 30 days (plus or minus 3 days) after surgery
food intake time | within the first 30 days (plus or minus 3 days) after surgery

SECONDARY OUTCOMES:
Complications | one year
readmission | one year